CLINICAL TRIAL: NCT02384122
Title: A Multicenter, Randomized, Open-label Clinical Trial Assessing the Efficacy of Octreotide in Decreasing Blood and Iron Requirements in Patients With Refractory Anemia Due to Angiodysplasias
Brief Title: Efficacy of Octreotide on Blood and Iron Requirements in Patients With Anemia Due to Angiodysplasias
Acronym: OCEAN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Jeroen Bosch Ziekenhuis (Other); Elisabeth-TweeSteden Ziekenhuis (Other); Catharina Ziekenhuis Eindhoven (Other); Bernhoven Hospital (Other); Tjongerschans hospital (Unknown); Gelre Hospitals (Other); Maasstad Hospital (Other); Reinier de Graaf Groep (Other); University Medical Center Groningen (Other); Rijnstate Hospital (Other); St. Antonius Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NLOCEAN.50514.091.14
Record Dates: First submitted 2015-03-04; First posted 2015-03-10 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-04

CONDITIONS: Angiodysplasia; Vascular Malformations; Gastrointestinal Hemorrhage; Anemia
Keywords: Angiodysplasias; Sandostatin LAR; Gastrointestinal bleeding; Somatostatin analogs; Octreotide
MeSH Terms: conditions — Angiodysplasia; Vascular Malformations; Gastrointestinal Hemorrhage; Anemia | interventions — Octreotide

STUDY DESIGN:
Intervention Model Description: Multicenter, open-label, randomized, parallel-group, superiority study to compare the efficacy of 40 mg octreotide long-acting release intramuscular every 28 days in addition to standard of care versus standard of care alone in patients with refractory anemia due to gastrointestinal bleeding from angiodysplasias.
Who Masked: Outcomes Assessor
Masking Description: The trial was blinded for the outcome adjudication committee but not for patients or attending physicians.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Octreotide (Active Comparator): Drug: Sandostatin LAR Sandostatin LAR 40 mg will be administered once every 4 weeks as a intramuscular injection
  Interventions: Drug: Octreotide
- Standard of care (No Intervention): Patients receive standard of care without a placebo.

INTERVENTIONS:
Drug: Octreotide — Two injections of 20 mg will be given monthly.
  Other Names: Sandostatin LAR; RVG 18236; ATC H01CB02
  Arms: Octreotide

SUMMARY:
The purpose of this study is to determine whether 40 mg octreotide long-acting release intramuscular every 28 days is effective in the treatment of patients with refractory anemia due to gastrointestinal angiodysplasias. We hypothesize that octreotide is effective in reducing the transfusion requirements (consisting of red blood cell transfusions and intravenous iron infusions) of patients with angiodysplasia-related anemia.

DETAILED DESCRIPTION:
Rationale: Gastrointestinal angiodysplasias are a common source of intractable small bowel bleeding, especially in older patients. Endoscopic ablation of angiodysplasias has limited efficacy and rebleeding rates are substantial. Recurrent bleeding results in refractory anemia which is managed with blood transfusions and/or iron infusions. Transfusion dependency reduces quality of life and is associated with substantial cardiovascular morbidity and mortality. Small cohort studies suggest a beneficial effect of octreotide in bleeding angiodysplasias, but evidence from rigorous, well-controlled studies are lacking.

Objective: To assess the efficacy of octreotide in reducing the transfusion requirements (consisting of blood transfusions and iron infusions) of patients with refractory anemia due to gastrointestinal angiodysplasias despite endoscopic intervention.

Study design: Multicenter, randomized, open-label intervention study.

Study population: Patients aged 18 years or older with transfusion-dependent anemia due to endoscopically confirmed angiodysplasias. Transfusion units consist of iron infusions (of 500 milligrams [mg]) and red blood cell (RBC) transfusions. At least one endoscopic attempt to treat the angiodysplasias needs to be recorded unless contra-indications are present. Patients with liver cirrhosis Child-Pugh C or liver failure, uncontrolled diabetes mellitus (defined by a glycated hemoglobin >64 mmol/mL), symptomatic cholecystolithiasis, and pregnant or nursing women, are regarded as ineligible because of the pharmacological profile of octreotide. Patients with hereditary hemorrhagic diseases or hematological disorders on active treatment, other alternative causes of gastrointestinal bleeding, presence of left ventricular assist devices, as well as patients with cancer under active treatment, and those with a life expectancy <1 year are excluded from enrolment

Intervention: Patients will be randomized (1:1) into two groups. The intervention group receives 40 mg octreotide long-acting release (Sandostatin LAR) every 28 days for a total period of 52 weeks as an adjunct to standard of care. The control group receives standard of care along. The last follow-up visit is in week 60.

Main study parameters/endpoints: The primary endpoint is defined as the mean difference in blood (RBC transfusions per 500 ml or packed cells) and parenteral iron (IV iron infusions per 500 mg) requirements between the intervention and control group, corrected for baseline transfusion requirements and follow-up time.

ELIGIBILITY:
Inclusion criteria:

* Endoscopically diagnosed angiodysplasias
* Transfusion dependency: at least 4 red blood cell transfusions (per 500 ml or packed cells) and/or parental iron infusions (per 500 mg) in the year before inclusion
* Failure of endoscopic therapy: at least one endoscopic attempt to coagulate the angiodysplasias or unsuitable for endoscopic procedures
* Providing informed consent
* Older than 18 years

Exclusion Criteria:

* Liver cirrhosis Child-Pugh C, liver failure or diagnosed portal hypertension
* Previous treatment with octreotide for the same indication (refractory anemia due to angiodysplasias)
* Current thalidomide treatment which is effective (no transfusion dependency)
* Life expectancy < 1 year
* Left ventricular assist devices (LVAD's)
* Hereditary hemorrhagic diseases or hematological disorders with active treatment
* Pregnancy or nursing women
* Uncontrolled diabetes as defined by HbA1C >64 mmol/ml, despite adequate therapy
* Known hypersensitivity to somatostatin analogs
* Symptomatic cholecystolithiasis
* Systemic cancer under active treatment (chemotherapy or radiation therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2022-07 (Actual); Study Completion 2023-05 (Actual)

PRIMARY OUTCOMES:
Difference in blood and parenteral iron requirements (transfusion units) | Study year (52 weeks)
  The mean difference in blood (RBC transfusions per 500 ml or packed cells) and parenteral iron (IV iron infusions per 500 mg) requirements between the intervention and standard of care arm, corrected for baseline transfusion requirements and follow-up time.

SECONDARY OUTCOMES:
Proportion with a good treatment response | During the study year (52 weeks) compared to the year (52 weeks) before randomization
  The proportion of patients in both groups that experienced a ≥50% (defined as a good response) and 100% (defined as a full response) reduction in the number of transfusion units received during the study year compared to baseline
Use of concomitant care | Study year (52 weeks)
  The proportion of patients in both groups that required concomitant care. Concomitant care consists of application of APC, discontinuation of antithrombotics, use of tranexamic acid, and starting octreotide in the control group.
Difference in endoscopic procedures | Study year (52 weeks)
  The mean difference in endoscopic procedures between both groups.
Difference in bleeding episodes | Study year (52 weeks)
  The mean difference in bleeding episodes between both groups. A bleeding episode is defined as each non-contiguous episode in which hospital care is sought for anemia.
Difference in healthcare utilization | Study year (52 weeks)
  The mean difference in healthcare utilization between both groups. Healthcare utilization consists of hospital admissions, ambulatory care, and emergency care.
Difference in hemoglobin levels | Study year (52 weeks)
  The mean difference in serum hemoglobin levels (mmol/L) between both groups.
Difference in ferritin levels | Study year (52 weeks)
  The mean difference in serum ferritin levels (ug/L) between both groups.
Difference in fatigue levels | Study year (52 weeks)
  The mean difference in fatigue levels between both groups. Fatigue is a patient-reported outcome measure (PROM), measured by the Multidimensional Fatigue Inventory (MFI-20), which covers five dimensions of fatigue affect and -tolerability. MFI-20 scores range from 20 (best) to 100 (worst).
Difference in quality of life | Study year (52 weeks)
  The mean difference in quality of life between both groups. Quality of life is a patient-reported outcome measure (PROM), measured by the Short Form Health Survey (SF-36), which uses eight subdomains to evaluate physical- and mental health. SF-36 scores range from 0 (worst) to 100 (best).
Difference in adverse events | Study year (52 weeks)
  The proportion of patients in both groups that experienced at least one adverse event (AE).
Difference in serious adverse events | Study year (52 weeks)
  The proportion of patients in both groups that experienced at least one serious adverse event (SAE).
Difference in mortality | Study year (52 weeks)
  The proportion of patients in both groups that died during the study.

OTHER OUTCOMES:
Subgroup analyses on blood transfusion dependency | Study year (52 weeks)
  Analyses include all patients that required at least one red blood cell transfusion (per 500 ml or packed cells) in the year before randomization (52 weeks).
Subgroup analyses on use of antithrombotics | Study year (52 weeks)
  Analyses include all patients that required at least one form of antithrombotics in the year before randomization (52 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Joost Drenth, MD. PhD, Principal Investigator — Radboud University Medical Center
Locations (12):
- Netherlands (12):
  - Gelre Hospital, Apeldoorn, Gelderland
  - Radboud University Medical Center (Radboudumc), Nijmegen, Gelderland
  - Jeroen Bosch Hospital, 's-Hertogenbosch, North Brabant
  - Catharina Hospital, Eindhoven, North Brabant
  - Elisabeth-TweeSteden Hospital, Tilburg, North Brabant
  - Reinier de Graaf Gasthuis, Delft, South Holland
  - St. Antonius Hospital, Nieuwegein, Utrecht
  - Rijnstate Hospital, Arnhem
  - University Medical Center Groningen (UMCG), Groningen
  - Tjongerschans Hospital, Heerenveen
  - Maasstad Hospital, Rotterdam
  - Bernhoven Hospital, Uden

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data and a data dictionary defining each field in the set will be available, upon reasonable request to Lia Goltstein and subjected to an appropriate data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Access Criteria: Data sharing agreement

REFERENCES:
- [Derived] Goltstein LCMJ, Grooteman KV, Bernts LHP, Scheffer RCH, Laheij RJF, Gilissen LPL, Schrauwen RWM, Talstra NC, Zuur AT, Braat H, Hadithi M, Brouwer JT, Nagengast WB, Oort FA, Tenthof van Noorden J, Kievit W, van Geenen EJM, Drenth JPH. Standard of Care Versus Octreotide in Angiodysplasia-Related Bleeding (the OCEAN Study): A Multicenter Randomized Controlled Trial. Gastroenterology. 2024 Apr;166(4):690-703. doi: 10.1053/j.gastro.2023.12.020. Epub 2023 Dec 28. PMID 38158089
- [Derived] Grooteman KV, van Geenen EJ, Drenth JP. Multicentre, open-label, randomised, parallel-group, superiority study to compare the efficacy of octreotide therapy 40 mg monthly versus standard of care in patients with refractory anaemia due to gastrointestinal bleeding from small bowel angiodysplasias: a protocol of the OCEAN trial. BMJ Open. 2016 Sep 12;6(9):e011442. doi: 10.1136/bmjopen-2016-011442. PMID 27619827
- See also: Announcement of research project in the "Nederlands Tijdschrift voor Geneeskunde" — https://www.ntvg.nl/system/files/publications/a8414.pdf
- Available data/document: Study Protocol: 27619827 — https://www.ncbi.nlm.nih.gov/pubmed/27619827